CLINICAL TRIAL: NCT03153371
Title: Early-onset Alzheimer's Disease Phenotypes: Neuropsychology and Neural Networks
Acronym: EOAD-Subtype
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Aging (NIA) (NIH); University of Southern California (Other)
Responsible Party: Principal Investigator, Mario F. Mendez, Professor of Neurology and Psychiatry, University of California, Los Angeles
Other Study IDs: 1RF1AG050967 (NIH); UCLA IRB#16-000496 (Other: UCLA Institutional Research Board); 1RF1AG050967-01A1 (NIH)
Record Dates: First submitted 2017-04-27; First posted 2017-05-15 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease, Early Onset; Alzheimer Disease; Alzheimer Disease, Late Onset; Dementia, Alzheimer Type; Logopenic Progressive Aphasia; Primary Progressive Aphasia; Visuospatial/Perceptual Abilities; Posterior Cortical Atrophy; Executive Dysfunction; Corticobasal Degeneration; Ideomotor Apraxia
Keywords: Alzheimer's disease; Young-onset; variant; visuospatial; language; apraxia; control; dementia; memory; MRI; neurology; neuropsychology; brain
MeSH Terms: conditions — Alzheimer Disease; Aphasia, Primary Progressive; Corticobasal Degeneration; Apraxia, Ideomotor; Language; Apraxias; Dementia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Early-onset Alzheimer's disease: This group will include 90 patients who have been diagnosed with clinically probable early-onset Alzheimer's disease by the UCLA Neurology Clinic (60 variant phenotypes; 30 typical amnestic).
- Alzheimer's disease: This group will include 30 patients who have been diagnosed with clinically probable Alzheimer's disease (typical late-onset AD)
- Controls: Healthy age-matched individuals without clinically significant cognitive impairments will be enrolled into this study.

SUMMARY:
This study attempts to identify two types of AD by using clinical and cognitive tasks and brain imaging. The subtypes of AD are separated into a "typical" group (memory loss) and a "variant" group (language, visuospatial, and other cognitive difficulties). Performance on the clinical tasks and brain imaging will be compared among the young-onset Alzheimer's disease group, a late-onset Alzheimer's disease group, and a control group.

DETAILED DESCRIPTION:
Unlike the usual late-onset Alzheimer's disease (LOAD), early-onset AD (EOAD), with onset before age 65, includes a high percentage of phenotypic variants. These non-familial, variants (vEOAD) present, not with progressive memory loss, but with language, visuospatial, or other cognitive difficulties. AD is now understood as a disorder that manifests with disturbed cognition reflecting disturbed neural networks. A multivariate analysis of neuropsychological tests, the "gold standard" for objectively defining neurocognitive impairments, coupled with structural and functional neuroimaging analysis of connectomes, can identify the neurocognitive-neural network profiles of vEOAD patients, compared to those with typical AD. This knowledge can increase our understanding of the heterogeneity of AD and how it causes disease.

This study hopes to show that vEOAD constitutes a "Type 2 AD", by (1) defining the neuropsychological components of Type 2 AD, and (2) understanding the anatomy and atrophy of the brains of vEOAD patients. Together, these components can outline the neurocognitive-neural network profile of Type 2 AD.

In addition to information that can help in the diagnosis and management of EOAD, this study can stimulate novel research into the reasons for this neurobiological heterogeneity in AD and could potentially lead to interventions based on alternate neurocognitive-neural network profiles.

ELIGIBILITY:
* Inclusion criteria for patients with Alzheimer's disease (AD):

  1. Meet criteria for AD.
  2. Meet clinical criteria for either typical amnestic AD or variant phenotypes of early-onset (EOAD, or "Type 2 AD").
  3. Mild-moderate dementia severity
  4. Sufficient English fluency to complete neuropsychological testing in English.
  5. Ability to provide consent for participation, or willingness to provide assent and a legally-authorized representative willing to provide surrogate consent.
  6. Availability of a caregiver informant for participation
* Exclusion criteria for patients with Alzheimer's disease (AD):

  1. Complicating medical illnesses.
  2. Significant primary visual impairments.
  3. Major psychiatric illness not due to the dementia.
  4. Confounding medications.
* Inclusion criteria for control participants:

  1. Score 28/30 or higher on the Folstein Mini-Mental Status Exam.
  2. Age 40-85 years old
  3. Able to provide consent for participation and express willingness to participate in one-year follow-up visits.
  4. Have sufficient English fluency to complete neuropsychological testing in English.
* Exclusion criteria for control participants:

  1. Complicating medical illnesses.
  2. Significant primary visual impairments.
  3. Major psychiatric illness not due to the dementia.
  4. Confounding medications.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of early-onset Alzheimer's disease (EOAD; with a diagnosis before age 65), including early-onset neurodegenerative conditions such as primary progressive aphasia (PPA), other aphasias (logopenic, semantic, and non-fluent), posterior cortical atrophy (PCA), ideomotor limb apraxias, and executive dysfunction.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2016-04-04 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Alzheimer's disease Subtype | Performed at baseline
  Neuropsychological testing results for use in a two-stage multivariate diagnostic method that combines the (weighted) test results in order to best discriminate Type 2 AD and typical AD.

SECONDARY OUTCOMES:
Change in overall Neurological profile | Performed at baseline and 1-year follow-up visit
  Change in performance on neurological tasks between baseline visit and follow-up visit.
Brain atrophy in MRI - Magnetic Resonance Imaging of the brain | Performed at baseline visit
  Images from initial MRI scan taken at baseline visit will be analyzed for atrophy and white matter tract integrity
Change in overall Neuropsychological profile | Performed at baseline and 1-year follow-up visit
  Change in neuropsychological performance over time.

CONTACTS AND LOCATIONS:
Overall Officials: Mario F Mendez, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Department of Neurology, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-12-19): https://cdn.clinicaltrials.gov/large-docs/71/NCT03153371/ICF_000.pdf